CLINICAL TRIAL: NCT03406598
Title: Impact of Bedside Visual Analysis of Sublingual Microcirculation in ICU Patients in Shock
Brief Title: Bedside Visual Analysis of Sublingual Microcirculation in Shock Patients
Acronym: MICROEYE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K170903J
Record Dates: First submitted 2017-12-20; First posted 2018-01-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Shock; Sepsis; Hemorrhagic Shock
Keywords: Shock; Microcirculation; Nurses
MeSH Terms: conditions — Shock; Sepsis; Shock, Hemorrhagic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in shock: Analysis of sublingual microcirculation by nurses in ICU patients in shock to predict needs for fluid challenge, vasopressors or transfusion.
  Interventions: Other: Patients in shock

INTERVENTIONS:
Other: Patients in shock — Analysis of sublingual microcirculation by nurses in ICU patients in shock to predict needs for fluid challenge, vasopressors or transfusion.

SUMMARY:
In shock patients, fluid resuscitation, infusion of vasopressors and transfusion are guided on hemodynamic macrovascular parameters. Analysis of sublingual microcirculation in shock patients is predictive of mortality and organ dysfunction. To optimize the quality of the resuscitation in shock patients, it could be useful to have an assessment of sublingual microcirculation in addition to the macrovascular parameters usually assessed by the nurses. But, this requires to have a monitor of sublingual microcirculation easy to use and to analyze at the bedside.

The primary outcome of the present study is to test the ability of visual analysis of sublingual microcirculation by nurses to predict needs for fluid challenge, vasopressors or transfusion in patients in shock. After ICU admission and study inclusion, the nurses in charge of the patient will perform a set of measurements of macrocirculatory and microcirculatory parameters every 4 h during the first three days after ICU admission and before and after every hemodynamic therapeutic intervention, such as fluid challenge, transfusion of red blood cells or change in catecholamine rate.

The secondary outcomes are to test 1/ to test the ability of visual analysis of sublingual microcirculation to predict organ dysfunction (SOFA score), and 2/ to evaluate the relationship between hemodynamic macrovascular and microvascular parameters. Intensive care patients in shock who need sedation, mechanical ventilation and invasive hemodynamic monitoring (Pulse Contour Cardiac Output (PiCCO 2 device)) will be included. In addition, patients will be included only when patients will obviously stay more than 24 hours in the ICU.

DETAILED DESCRIPTION:
In shock patients, fluid resuscitation, infusion of vasopressors and transfusion are guided on hemodynamic macrovascular parameters as arterial pressure, cardiac output, lactate and diuresis. Analysis of sublingual microcirculation in shock patients is predictive of mortality and organ dysfunction. To optimize the quality of the resuscitation in shock patients, it could be useful to have an assessment of sublingual microcirculation in addition to the macrovascular parameters usually assessed by the nurses. But, this requires to have a monitor of sublingual microcirculation easy to use and to analyze at the bedside. In a previous study, using a side-stream dark-field (SDF) imaging device (Cytocam video microscope, Braedius®, Netherlands), the investigators have reported that a real-time nurse bedside qualitative evaluation of Microvascular flow index (MFI) had a good agreement with conventional delayed physician analysis, and was highly sensitive and specific for detecting impaired microvascular flow and low capillary density.

The primary outcome of the present study is to test the ability of visual analysis of sublingual microcirculation by nurses in patients in shock to predict needs for fluid challenge, vasopressors or transfusion.

The secondary outcomes are:

1. To test the ability of visual analysis of sublingual microcirculation to predict organ dysfunction (SOFA score)
2. To evaluate the relationship between hemodynamic macrovascular and microvascular parameters. The investigators will consider the macrovascular parameters usually collected by nurses each 4h: arterial pressure, heart rate, cardiac index, stroke volume index, global end-diastolic blood volume, extravascular lung water, the respiratory variations of pulse pressure (delta PP), lactate, hemoglobin, venous-to-arterial carbon dioxide differences (Pv-aCO2), diuresis and the microvascular parameters (MFI and capillary density).

Study design and measurements After ICU admission and study inclusion, the nurses in charge of the patient will perform a set of measurements of macrocirculatory and microcirculatory parameters every 4 h during the first three days after ICU admission and before and after every hemodynamic therapeutic intervention, such as fluid challenge, transfusion of red blood cells or change in catecholamine rate during this period.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care patients in shock who need sedation, mechanical ventilation and invasive hemodynamic monitoring (Pulse Contour Cardiac Output (PiCCO 2 device)).
* In addition, patients will be included only when patients will obviously stay more than 24 hours in the ICU.

Exclusion Criteria:

* Maxillofacial trauma
* Oral mucosal injuries preventing to perform the sublingual microcirculation monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive care patients in shock who need sedation, mechanical ventilation and invasive hemodynamic monitoring (Pulse Contour Cardiac Output (PiCCO 2 device)).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-03-02 (Actual); Primary Completion 2021-10-10 (Estimated); Study Completion 2021-10-10 (Estimated)

PRIMARY OUTCOMES:
Measured of Microvascular Flow Index (MFI) | Every 4 hours during 3 days
  Each set of measurements will consist of three successive video sequences of 20 seconds at three different sites. The nurse will calculate the MFI score. The image will be divided into 4 quadrants and the vessels <20 μm diameter will be assigned a score based on the predominant flow characteristics of the vessels in that quadrant (0 = absent flow; 1 = intermittent; 2 = sluggish; 3 = normal). The values in each quadrant are averaged to give an MFI score for each sublingual site at each time point

SECONDARY OUTCOMES:
SOFA score | Every 4 hours during 3 days
  To test the ability of visual analysis of sublingual microcirculation to predict organ dysfunction
Hemodynamic macrovascular parameters | Every 4 hours during 3 days
  To evaluate the relationship between hemodynamic macrovascular and microvascular parameters. We will consider the macrovascular parameters usually collected by nurses each 4h: arterial pressure, heart rate, cardiac index, stroke volume index, global end-diastolic blood volume, extravascular lung water, the respiratory variations of pulse pressure (delta PP), lactate, hemoglobin, venous-to-arterial carbon dioxide differences (Pv-aCO2), diuresis and the microvascular parameters (MFI and capillary density)
Hemodynamic microvascular parameters. | Every 4 hours during 3 days
  To evaluate the relationship between hemodynamic macrovascular and microvascular parameters. We will consider the macrovascular parameters usually collected by nurses each 4h: arterial pressure, heart rate, cardiac index, stroke volume index, global end-diastolic blood volume, extravascular lung water, the respiratory variations of pulse pressure (delta PP), lactate, hemoglobin, venous-to-arterial carbon dioxide differences (Pv-aCO2), diuresis and the microvascular parameters (MFI and capillary density)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques DURANTEAU, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Département d'Anesthésie Réanimation, Le Kremlin-Bicêtre, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Backer D, Donadello K, Sakr Y, Ospina-Tascon G, Salgado D, Scolletta S, Vincent JL. Microcirculatory alterations in patients with severe sepsis: impact of time of assessment and relationship with outcome. Crit Care Med. 2013 Mar;41(3):791-9. doi: 10.1097/CCM.0b013e3182742e8b. PMID 23318492
- [Background] Tachon G, Harrois A, Tanaka S, Kato H, Huet O, Pottecher J, Vicaut E, Duranteau J. Microcirculatory alterations in traumatic hemorrhagic shock. Crit Care Med. 2014 Jun;42(6):1433-41. doi: 10.1097/CCM.0000000000000223. PMID 24561562
- [Background] Tanaka S, Harrois A, Nicolai C, Flores M, Hamada S, Vicaut E, Duranteau J. Qualitative real-time analysis by nurses of sublingual microcirculation in intensive care unit: the MICRONURSE study. Crit Care. 2015 Nov 6;19:388. doi: 10.1186/s13054-015-1106-3. PMID 26542952
- [Background] Massey MJ, Larochelle E, Najarro G, Karmacharla A, Arnold R, Trzeciak S, Angus DC, Shapiro NI. The microcirculation image quality score: development and preliminary evaluation of a proposed approach to grading quality of image acquisition for bedside videomicroscopy. J Crit Care. 2013 Dec;28(6):913-7. doi: 10.1016/j.jcrc.2013.06.015. Epub 2013 Aug 21. PMID 23972316